CLINICAL TRIAL: NCT01325506
Title: Effectiveness of Open and Robotic Prostatectomy: The PROSTQA-RP2 Study
Brief Title: Effectiveness of Open and Robotic Prostatectomy
Acronym: PROSTQA-RP2
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); The Cleveland Clinic (Other); Johns Hopkins University (Other); University of California, San Francisco (Other); University of Michigan (Other); Vanderbilt University (Other); Washington University School of Medicine (Other); Emory University (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter Chang, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 10-155
Record Dates: First submitted 2011-03-09; First posted 2011-03-29 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prostatectomy subjects
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire, telephone interviews, and clinical follow-up

SUMMARY:
Prostate cancer is the most common cancer in American men. Surgical removal of the entire prostate (prostatectomy) is one option among the various ways to treat prostate cancer. The use of robot assistance for prostatectomy has become common place, but its effectiveness has not been compared to standard open prostatectomy in trials carried out at more than one medical institution in which participants are identified and followed forward in time. Robot assisted and standard open prostatectomy health related quality of life (HRQOL) outcomes have not been compared in a prospective, multi-centered study. Prostatectomy can have side effects that can change with time. This research study seeks to determine how common and how long-lasting such side effects are; to find out what features of individual men's cancers and what features of the treatments affect those side effects. This study also seeks to identify factors that affect the quality of prostate cancer care by looking at how satisfied men are with their prostate cancer care. Through these findings, this study aims to allow treatment side effects to be anticipated more accurately for individual patients, and to provide a means for determining the quality of prostate care.

DETAILED DESCRIPTION:
The investigators will follow your prostate cancer treatment outcomes and health related quality of life following prostatectomy by asking you direct questions, collect information from medical records and phone interviews.

Information about your prostate cancer treatment, and related health concerns, and information regarding the cost of care, may also be collected from your medical record, other medical center sources, and your primary care provider (PCP). Clinical information will be collected: prior to beginning treatment (prostatectomy); 6 month, 12 months, 18 months, and 24 months after your prostatectomy; once a year thereafter for possibly up to 12 years.

You will be asked to take part in six telephone interviews regarding quality of life, possible therapy side effects, and satisfaction with prostate cancer therapy. Each phone interview should last 15-25 minutes. All questions are voluntary. The phone interviews will be conducted: prior to beginning treatment (prostatectomy); 2 months, 6 months, 12 months, 18 months, and 24 months after prostatectomy; 10 additional phone interviews may be conducted (once a year thereafter, for possibly up to 12 years).

ELIGIBILITY:
Inclusion Criteria:

* Early stage prostate cancer (AJCC [2002] clinical stage < or = T2NXMX; T stage is based on rectal exam findings alone).
* Gleason score based on local pathology within 12 months of registration. (Patients with an original diagnosis of prostate cancer proceeding 12 months are also eligible but pathology confirmation of cancer within 12 months of registration is required.)
* Serum PSA test result from within 12 months of registration
* Able to participate in baseline and follow-up phone interviews conducted in English
* Scheduled to undergo Open Radical Prostatectomy or Robotic Assisted Laparoscopic Prostatectomy

Exclusion Criteria:

* Previous definitive primary prostate cancer therapy (prostatectomy, external radiation, brachytherapy, cryotherapy, or other interventions)
* Previous radiation therapy to the pelvis
* Previous major reconstructive or extirpative pelvic surgery (including but not limited to abdominal-perineal resection, or penile implant)
* Previous androgen suppression therapy (LHrH agonist or antagonist), anti-androgen therapy (Casodex, Flutamide, or Nilandron), or estrogen therapy (DES or PC-SPEZ). (Prior or current finasteride or dutasteride therapy is allowed)
* Known urethral stricture
* Urostomy or colostomy
* Chronic urinary catheterization

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with localized prostate cancer who have elected to undergo a robot assisted laparoscopic prostatectomy or an open prostatectomy from participating clinical sites
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2010-09; Primary Completion 2024-10 (Actual); Study Completion 2024-10 (Actual)

PRIMARY OUTCOMES:
To compare clinical outcomes between robot assisted laparoscopic prostatectomy (RALP) and open retropubic prostatectomy (ORP). | Eligible participants will initially be followed for 2 years with the possibility for up to 12 years.
  Outcomes include: acute clinical morbidity (thromboembolic events, bleeding requiring transfusion, surgical infection, other events requiring intervention within 30 days of prostatectomy) and satisfaction with overall treatment outcome; cancer control (surgical margins, PSA recurrence-free survival, requirement of salvage or adjuvant treatment).
To compare patient-reported outcomes between robot assisted laparoscopic prostatectomy (RALP) and open retropubic prostatectomy (ORP). | Eligible participants will initially be followed for 2 years with the possibility for up to 12 years.
  Outcomes include: patient-reported outcomes (urinary incontinence, erectile dysfunction) and satisfaction with overall treatment outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sanda, MD, Principal Investigator — Emory Healthcare; Peter Chang, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - Emory Healthcare, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University Medical Center St. Louis, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Chang P, Wagner AA, Regan MM, Smith JA, Saigal CS, Litwin MS, Hu JC, Cooperberg MR, Carroll PR, Klein EA, Kibel AS, Andriole GL, Han M, Partin AW, Wood DP, Crociani CM, Greenfield TK, Patil D, Hembroff LA, Davis K, Stork L, Spratt DE, Wei JT, Sanda MG; PROST-QA/RP2 Consortium. Prospective Multicenter Comparison of Open and Robotic Radical Prostatectomy: The PROST-QA/RP2 Consortium. J Urol. 2022 Jan;207(1):127-136. doi: 10.1097/JU.0000000000002176. Epub 2021 Aug 26. PMID 34433304